CLINICAL TRIAL: NCT01609933
Title: An Open-Label Study to Evaluate the Safety, Antiviral Activity and Pharmacokinetics of Direct-Acting Antiviral Agent (DAA) Treatment in Combination With Peginterferon Alpha-2a and Ribavirin (pegIFN/RBV) in Chronic Hepatitis C Virus (HCV) Infected Subjects Who Have Experienced Virologic Failure in a Previous AbbVie or Abbott DAA Combination Study
Brief Title: A Study to Evaluate the Safety and Effect of Treatment With Experimental Antiviral Drugs in Combination With Peginterferon Alpha-2a and Ribavirin in People With Hepatitis C Virus Who Did Not Respond to Treatment in a Previous AbbVie/Abbott Combination Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AbbVie (prior sponsor, Abbott) (Industry)
Responsible Party: Sponsor
Organization: AbbVie (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M13-101
Record Dates: First submitted 2012-05-30; First posted 2012-06-01 (Estimated); Results first posted 2018-06-19 (Actual); Last update posted 2018-06-19 (Actual); Status verified 2018-05

CONDITIONS: Chronic Hepatitis C
Keywords: Hepatitis C Virus (HCV); Hepatitis C Genotype 1; Chronic Hepatitis C; HCV
MeSH Terms: conditions — Hepatitis C, Chronic; Hepatitis C | interventions — paritaprevir; Ritonavir; ombitasvir; peginterferon alfa-2a; Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- 2-DAA + PegIFN/RBV (Experimental): 2-direct-acting antiviral (2-DAA: ABT-450 [paritaprevir] 200 mg once daily [QD], ritonavir 100 mg QD, ABT-267 [ombitasvir] 25 mg QD) plus pegylated interferon alpha-2a (pegIFN) 180 mcg once weekly and Ribavirin (RBV) weight-based dosing, 1000 to 1200 mg divided twice daily (BID) for 24 weeks (Substudy 1) and followed by pegIFN and RBV alone for an additional 24 weeks (Substudy 2).
  Interventions: Drug: ABT-450/r; Drug: ABT-267; Drug: pegylated interferon alpha-2a (pegIFN); Drug: Ribavirin (RBV)

INTERVENTIONS:
Drug: ABT-450/r — ABT-450 (tablets) dosed with ritonavir (capsules or tablets)
  Other Names: ABT-450 also known as paritaprevir and r is also know as ritonavir
Drug: ABT-267 — ABT-267 (tablets)
  Other Names: ABT-267 also known as ombitasvir
Drug: pegylated interferon alpha-2a (pegIFN) — pegIFN alpha-2a (syringe)
Drug: Ribavirin (RBV) — Ribavirin (tablets)

SUMMARY:
A study to evaluate the safety and effect of treatment with experimental antiviral drugs in combination with peginterferon alpha-2a and ribavirin in people with hepatitis C virus who did not respond to treatment in a previous AbbVie/Abbott combination study.

ELIGIBILITY:
Inclusion Criteria:

Main Inclusion: To be enrolled in this protocol, subjects must meet all of the following inclusion criteria:

* Subject must have experienced virologic failure as defined in a previous AbbVie/Abbott direct-acting antiviral (DAA) combination trial.
* Female subjects of childbearing potential must be willing to use two effective forms of birth control (not including oral contraceptives or contraceptives containing ethinyl estradiol) while receiving study drug and for 7 months (or per local ribavirin label) after stopping study drug.
* Males must be surgically sterile or have male partners only or agree to practice two effective forms of birth control throughout the course of the study, starting with Study Day 1 and for 7 months (or per local ribavirin label) after the last dose of study drug, unless abstinent from sexual intercourse.
* Subject must be considered an appropriate candidate for peginterferon (pegIFN) alpha-2a, ribavirin (RBV), ABT-450/ritonavir (r) and ABT-267 therapy in the opinion of the investigator.
* Subject is infected with hepatitis C virus (HCV) genotype 1 at screening.

Subjects diagnosed with cirrhosis must also meet the following criteria:

* Compensated cirrhosis defined as Child-Pugh score of ≤ 6 at Screening.
* Absence of hepatocellular carcinoma based on a negative ultrasound, computed tomography (CT) scan or magnetic resonance imaging (MRI) performed within 3 months prior to Screening or during the Screening period.

Exclusion Criteria:

* In subjects with a prior null or partial response to pegIFN/RBV treatment at any time prior to pre-screening for this study or any prior failure with pegIFN/RBV plus telaprevir, the presence of variants relative to the appropriate prototypic reference sequence (H77 for 1a or Con1 for 1b) at any of the following positions: NS3 155, 156, or 168; or NS5A 28, 29, 30, 31, 32, 58, or 93.
* Females who are pregnant or plan to become pregnant, or breast-feeding, or males whose partners are pregnant or planning to become pregnant within 7 months (or per local RBV label) after their last dose of RBV.
* Use of known strong inducers (e.g., phenobarbital, rifampin, carbamazepine, St. John's Wort) of Cytochrome P450 3A (CYP3A) within 2 weeks prior to study drug administration.
* Use of any medications contraindicated for use with pegIFN alpha-2a, RBV or ritonavir within 2 weeks prior to study drug administration. Prior to entering the study, subjects must be able to safely discontinue the contraindicated medication or switch to an acceptable alternative under supervision of the investigator.
* Discontinuation of antiviral therapy due to intolerance or a DAA- or RBV-associated adverse event in a previous AbbVie/Abbott DAA combination study.

Subjects with compensated cirrhosis must also not meet the following criteria:

* Any current or past clinical evidence of Child-Pugh B or C Classification or clinical history of liver decompensation such as ascites (noted on physical exam), variceal bleeding or hepatic encephalopathy.
* Serum Alpha-Fetoprotein (sAFP) > 100 ng/mL at Screening.
* A screening ultrasound suspicious for hepatocellular carcinoma and confirmed with a subsequent CT scan or MRI during the screening period.

Ages: 18 Years to 71 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2012-12-18 (Actual); Primary Completion 2017-05-03 (Actual); Study Completion 2017-05-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: AbbVie Inc., Study Director — AbbVie

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Bernstein D, Tripathi R, Cohen DE. Ombitasvir, paritaprevir, and ritonavir with peginterferon-alpha2a plus ribavirin in treatment-experienced patients with chronic hepatitis C virus genotype 1 infection. Hepat Med. 2019 Feb 13;11:35-40. doi: 10.2147/HMER.S189158. eCollection 2019. PMID 30858739

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study included a 42-day screening period.
Groups:
- 2-DAA + PegIFN/RBV: 2-direct-acting antiviral (2-DAA: ABT-450 [paritaprevir] 200 mg once daily [QD], ritonavir 100 mg QD, ABT-267 [ombitasvir] 25 mg QD) plus pegylated interferon alpha-2a (pegIFN) 180 mcg once weekly and Ribavirin (RBV) weight-based dosing, 1000 to 1200 mg divided twice daily (BID) for 24 weeks and followed by pegIFN and RBV alone for an additional 24 weeks.
Period: Overall Study
Arm/Group | 2-DAA + PegIFN/RBV
Started | 32
Completed | 28
Not Completed | 4
Not completed — Adverse Event | 1
Not completed — Withdrawal by Subject | 3

BASELINE CHARACTERISTICS:
Population: All subjects who received at least 1 dose of study drug were included in the intent-to-treat (ITT) population; the safety population is the same as the ITT population.
Arm/Group | 2-DAA + PegIFN/RBV
Number analyzed (Participants) | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.4 (9.77)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 25
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 30
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving Sustained Virologic Response 12 Weeks Post Treatment (SVR12)
Description: SVR12 was defined as hepatitis C virus ribonucleic acid (HCV RNA) level less than lower limit of quantitation [LLOQ] 12 weeks after the last dose of study drugs (DAAs plus pegIFN alpha-2a and RBV).
Time Frame: 12 weeks after last dose of study drugs (DAAs plus pegIFN alpha-2a and RBV); approximately 36 weeks after subject's initial dose of study drug in Substudy 1
Population: ITT population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- 2-DAA + PegIFN/RBV: 2-direct-acting antiviral (2-DAA: ABT-450 [paritaprevir] 200 mg once daily [QD], ritonavir 100 mg QD, ABT-267 [ombitasvir] 25 mg QD) plus pegylated interferon alpha-2a (pegIFN) 180 mcg once weekly and Ribavirin (RBV) weight-based dosing, 1000 to 1200 mg divided twice daily (BID) for 24 weeks followed by pegIFN and RBV alone for an additional 24 weeks.
Arm/Group | 2-DAA + PegIFN/RBV
Number analyzed (Participants) | 32
percentage of participants | 81.3 [64.7 to 91.1]

2. Secondary Outcome: Percentage of Participants Achieving Virologic Response 24 Weeks Post Treatment (SVR24)
Description: SVR24 was defined as HCV RNA level less than the LLOQ 24 weeks after the last dose of study drugs (DAAs plus pegIFN alpha-2a and RBV).
Time Frame: 24 weeks after last dose of study drugs (DAAs plus pegIFN alpha-2a and RBV); approximately 48 weeks after subject's initial dose of study drug in Substudy 1
Population: ITT population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 2-DAA + PegIFN/RBV
Number analyzed (Participants) | 32
percentage of participants | 78.1 [61.2 to 89.0]

3. Secondary Outcome: Percentage of Participants With Extended Rapid Virologic Response (eRVR)
Description: eRVR was defined as HCV RNA level < LLOQ at Substudy 1 treatment weeks 4 through 12 without a confirmed HCV RNA >= LLOQ
Time Frame: Treatment weeks 4 through 12 of Substudy 1 (DAAs plus pegIFN alpha-2a and RBV)
Population: ITT Population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 2-DAA + PegIFN/RBV
Number analyzed (Participants) | 32
percentage of participants | 87.5 [71.9 to 95.0]

4. Secondary Outcome: Number of Participants With Adverse Events
Description: An adverse event (AE) is defined as any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment. The investigator assessed the relationship of each event to the use of study drug as either probably related, possibly related, probably not related or not related. A serious adverse event (SAE) is an event that results in death, is life-threatening, requires or prolongs hospitalization, results in a congenital anomaly, persistent or significant disability/incapacity or is an important medical event that, based on medical judgment, may jeopardize the subject and may require medical or surgical intervention to prevent any of the outcomes listed above. Treatment-emergent events (TEAEs/TESAEs) are defined as any event that began or worsened in severity after initiation of study drug through 30 days post-DAA dosing. For more details on AEs, see the AE section.
Time Frame: From first dose of study drug through 30 days after last dose of study drug (DAAs plus pegIFN alpha-2a and RBV) (up to 28 weeks).
Population: Safety population (all subjects who received at least 1 dose of study drug)
Measure: Number; unit: participants
Groups:
- 2-DAA + PegIFN/RBV: 2-direct-acting antiviral (2-DAA: ABT-450 [paritaprevir] 200 mg once daily [QD], ritonavir 100 mg QD, ABT-267 [ombitasvir] 25 mg QD) plus pegylated interferon alpha-2a (pegIFN) 180 mcg once weekly and Ribavirin (RBV) weight-based dosing, 1000 to 1200 mg divided twice daily (BID).
Arm/Group | 2-DAA + PegIFN/RBV
Number analyzed (Participants) | 32
participants
  2-DAA TEAE | 29
  2-DAA TESAE | 1

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events (TEAEs) and serious adverse events (TESAEs) were collected from first dose of study drug through 30 days after the last dose of DAA (2-DAA + pegIFN alpha-2a and RBV) dosing (up to 28 weeks).
Description: TEAEs and TESAEs are defined as any AE with an onset date that is after the first dose of study drug through 30 days after the last dose of DAAs (up to 28 weeks) and were collected whether elicited or spontaneously reported by the participant.
Arm/Group | 2-DAA + PegIFN/RBV
All-Cause Mortality (participants affected / at risk) | 1/32
Serious Adverse Events (participants affected / at risk) | 1/32
Other Adverse Events (participants affected / at risk) | 28/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 2-DAA + PegIFN/RBV (N=32)
MYOCARDIAL INFARCTION (Cardiac disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 2-DAA + PegIFN/RBV (N=32)
LYMPHOPENIA (Blood and lymphatic system disorders) | 2 (2)
NEUTROPENIA (Blood and lymphatic system disorders) | 7 (10)
VISION BLURRED (Eye disorders) | 2 (3)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 3 (3)
ANAL PRURITUS (Gastrointestinal disorders) | 2 (2)
DIARRHOEA (Gastrointestinal disorders) | 6 (7)
DRY MOUTH (Gastrointestinal disorders) | 2 (2)
NAUSEA (Gastrointestinal disorders) | 9 (9)
ASTHENIA (General disorders) | 2 (2)
CHILLS (General disorders) | 3 (3)
FATIGUE (General disorders) | 11 (13)
FEELING ABNORMAL (General disorders) | 2 (2)
INFLUENZA LIKE ILLNESS (General disorders) | 6 (6)
PAIN (General disorders) | 3 (4)
PYREXIA (General disorders) | 4 (4)
JAUNDICE (Hepatobiliary disorders) | 2 (2)
BRONCHITIS (Infections and infestations) | 2 (3)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 3 (3)
VIRAL INFECTION (Infections and infestations) | 2 (2)
VIRAL UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 2 (2)
NEUTROPHIL COUNT DECREASED (Investigations) | 3 (7)
WEIGHT DECREASED (Investigations) | 2 (2)
WHITE BLOOD CELL COUNT DECREASED (Investigations) | 5 (7)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 2 (2)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 3 (4)
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 2 (2)
MYALGIA (Musculoskeletal and connective tissue disorders) | 2 (2)
DISTURBANCE IN ATTENTION (Nervous system disorders) | 3 (3)
HEADACHE (Nervous system disorders) | 14 (27)
ANXIETY (Psychiatric disorders) | 2 (2)
DEPRESSION (Psychiatric disorders) | 2 (2)
INSOMNIA (Psychiatric disorders) | 8 (10)
IRRITABILITY (Psychiatric disorders) | 4 (4)
COUGH (Respiratory, thoracic and mediastinal disorders) | 4 (4)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 4 (4)
DRY SKIN (Skin and subcutaneous tissue disorders) | 4 (6)
PRURITUS (Skin and subcutaneous tissue disorders) | 6 (8)
RASH (Skin and subcutaneous tissue disorders) | 8 (9)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Study Protocol (2015-06-26): https://cdn.clinicaltrials.gov/large-docs/33/NCT01609933/Prot_000.pdf
  • Statistical Analysis Plan (2017-05-05): https://cdn.clinicaltrials.gov/large-docs/33/NCT01609933/SAP_001.pdf